CLINICAL TRIAL: NCT02720887
Title: Single-center Prospective Descriptive Study Evaluating the Presence of Nanoparticles in the Amniotic Fluid in Pregnant Women
Brief Title: Presence of Nanoparticles in the Amniotic Fluid
Acronym: NAMIOTIC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: SAINBIOSE (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1608016; 2016-A00250-51 (Other: ANSM)
Record Dates: First submitted 2016-03-11; First posted 2016-03-28 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Intrauterine Disorder
Keywords: pregnant women; nanoparticles; amniotic fluid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — amniotic fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant woman: Patient to receive an amniocentesis for medical reasons other than study and who will have a measure of nanoparticles load
  Interventions: Procedure: Nanoparticles load

INTERVENTIONS:
Procedure: Nanoparticles load — Pregnant women will have a sampling of amniotic fluid to measure load and composition of nanoparticles.

SUMMARY:
The nanoparticles (NP) are defined as particles whose size is no greater than 100 nanometers. However, their impact on health remains little evaluated.

Placental transfer of NP has been proven in many studies in vitro and in vivo in animals, and toxicity in the fetus has been studied in many animals. The investigators seem interesting at first to establish the mineralogical load in the amniotic fluid in humans.

The first objective of this study is to determine the mineralogical NP load, quantity and composition, in the amniotic fluid in pregnant women.

DETAILED DESCRIPTION:
The analysis will be done on 100 amniotic fluid samples and 100 blood samples. Particle size analysis will be performed by a technique of dynamic light scattering, which permits the distribution by volume or by number of NP according to their size. Parallel to the different chemical species present in the sample must be measured by atomic emission spectrometry with inductively coupled plasma.

The results of this study will be useful for further studies on the fetal toxicity of NP in humans.

ELIGIBILITY:
Inclusion Criteria:

* Patient major
* Patient to receive an amniocentesis for medical reasons other than study (serum marker of the first quarter with an increased risk of trisomy 21 greater than 1/250, amniodrainage, sonographic sign of call)
* Patient who have given their free, informed and signed

Exclusion Criteria:

* Inability to make withdrawals

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women who receive an amniocentesis for medical reasons other than study
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Percentage of nanoparticles in amniotic fluid (%) | day 1
  Percentage of each mineralogical Nanoparticle present in the amniotic fluid

SECONDARY OUTCOMES:
Percentage of nanoparticles in blood | day 1
  Percentage of each mineralogical Nanoparticle present in maternal blood
Correlation Nanoparticles between blood and amniotic fluid | day 1
  Establish a correlation between the mineralogical NP load in amniotic fluid and maternal blood.

CONTACTS AND LOCATIONS:
Overall Officials: Celine CHAULEUR, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raia-Barjat T, Prieux C, Leclerc L, Sarry G, Grimal L, Chauleur C, Pourchez J, Forest V. Elemental fingerprint of human amniotic fluids and relationship with potential sources of maternal exposure. J Trace Elem Med Biol. 2020 Jul;60:126477. doi: 10.1016/j.jtemb.2020.126477. Epub 2020 Feb 27. PMID 32142960